CLINICAL TRIAL: NCT05739994
Title: Frontal and Parietal Contributions to Proprioception and Motor Skill Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Hannah Justine Block, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17096; R01NS112367-01A1 (NIH)
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Basic Science

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dorsolateral prefrontal cortex (DLPFC) (Experimental): Theta burst transcranial magnetic stimulation (cTBS) will be applied over dorsolateral prefrontal cortex (DLPFC).
  Interventions: Other: Theta burst transcranial magnetic stimulation
- Supramarginal gyrus (SMG) (Experimental): Theta burst transcranial magnetic stimulation (cTBS) will be applied over the supramarginal gyrus (SMG).
  Interventions: Other: Theta burst transcranial magnetic stimulation
- Sham control group (Sham Comparator): Sham theta burst transcranial magnetic stimulation (cTBS) will be applied over the vertex.
  Interventions: Other: Sham theta burst transcranial magnetic stimulation

INTERVENTIONS:
Other: Theta burst transcranial magnetic stimulation — Continuous theta burst TMS (cTBS) will be delivered to a location on the head. cTBS consists of 600 low-intensity TMS pulses delivered over 40 seconds in a pattern of 50 Hz triplets delivered at 5 Hz.
  Arms: Dorsolateral prefrontal cortex (DLPFC); Supramarginal gyrus (SMG)
Other: Sham theta burst transcranial magnetic stimulation — Continuous theta burst TMS (cTBS) will be delivered near the head, while an unplugged TMS coil is held at the vertex. No current will be induced in the head with this procedure.
  Arms: Sham control group

SUMMARY:
The purpose of this study is to understand how the different regions of the brain affect our sense of limbs in space (proprioception) and in turn our hand movements (motor skill learning). This information might help us one day to generate better rehabilitation protocols to help patients with movement deficits.

DETAILED DESCRIPTION:
Moving our hands accurately, and learning new movement skills, depends on accurate sensory information. One of the sensory inputs which is crucial to make accurate movements is proprioception (sense of our limbs in space). Failure in estimating hand position results in inaccurate movement, raising the potential for accidents and injuries, but how the healthy brain carries out these functions, and how they could be strengthened in populations with sensory and motor deficits (e.g. stroke), is unknown. With greater understanding of these processes in the healthy brain, it may one day be possible to develop rehabilitation strategies that target a patient's unique mix of sensory and motor deficits.

A robust way to identify whether a brain region plays a role in a behavior is to temporarily modulate its excitability in healthy people using non-invasive brain stimulation. This is commonly done in research with a short sequence of low-intensity transcranial magnetic stimulation (TMS), also known as repetitive TMS (rTMS). rTMS is used clinically to treat conditions such as depression and is considered very low risk provided the generally accepted screening criteria are met. In the research setting, this technique is widely used not only in healthy adults (as in this study) but also in children and people with concussion, stroke, Parkinson's disease, and more.

In separate groups of subjects, we will use rTMS over one of several brain regions of interest before the subject In separate groups of subjects, we will use a 40-second sequence of rTMS called continuous theta burst stimulation (cTBS) over one of several brain regions of interest before the subject performs performs proprioceptive and skill learning tasks known to involve sensory and motor skill (learning). If performance of the task is affected by rTMS for a given group (relative to the sham, or control, group), it means that brain region plays some role in that type of proprioceptive or skill task.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must be between the ages of 18-45 years old and right-handed.
* We will only test right-handed individuals.
* We will only include individuals who report being free of Covid symptoms in week preceding testing.

Exclusion Criteria:

* Current vision problems, other than needing glasses or contacts.
* Subjects will also be excluded if they currently suffer from frequent severe headaches, glaucoma, heart or respiratory disease, hypertension, psychiatric conditions, or learning or attention conditions.
* They will also be excluded for current or past: visual, hearing, or balance impairments; stroke, seizure/epilepsy (including family history), or severe head trauma; fainting; or diabetes.
* Subjects will be excluded for metal implants in the head other than titanium; cochlear implants; implanted neurostimulator; cardiac pacemaker; intracardiac lines; or a medication infusion device.
* Because TMS does not penetrate deeply into the head, we cannot test subjects whose hair does not permit contact between the TMS coil and the scalp. We will therefore exclude subjects with dreadlocks, weaves, or hair extensions.
* To protect the data from extraneous peripheral influences, we will also exclude subjects who have had serious injury to the bones, joints, or muscles of either hand or arm, and have not fully recovered. For the purpose of this study, "fully recovered" means they no longer notice any pain, weakness, or loss of sensation in the injured area, and have no mobility limitations.
* For the validity of our data, we will exclude subjects taking medications or drugs that are known to affect cortical excitability and possibly seizure risk in an rTMS study. These medications/drugs are (Rossi et al., 2009): imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), theophylline, mianserin, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, reboxetine, venlafaxine, duloxetine, bupropion, mirtazapine, fluphenazine, pimozide, haloperidol, olanzapine, quetiapine, aripiprazole, ziprasidone, risperidone, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporin, chlorambucil, vincristine, methotrexate, cytosine arabinoside, BCNU, lithium, anticholinergics, antihistamines, sympathomimetics.
* Participants will also be excluded if they have metallic, mechanical, or magnetic implants; are claustrophobic, or are unable to remain still for long periods of time; or use an intra-uterine device (IUD) whos MR compatibility has not been established.
* Women who are pregnant or think they might be pregnant will also be excluded, as effects of fMRI on the unborn are not known.
* People who have a BMI over 30 will be excluded as it may be uncomfortable or impossible to lay in the MRI scanner.
* Potential subjects will be invited to reschedule if they would otherwise be eligible (according to the initial screening), but the day of testing have drunk more than 3 units of alcohol or taken other recreational drugs in the 24 hour period prior to testing; have had more than 3 cups of coffee in the last hour; are sleep deprived (<4 hours sleep the previous night); or have participated in another brain stimulation experiment the same day. These are standard in the TMS literature to protect the validity of the data and keep seizure risk minimal. In addition, we will invite invite subjects to reschedule if they have any of the common Covid symptoms within the last week. If they don't believe they can meet these criteria on another date, they will be excluded.
* After giving their consent, participants may be excluded during or after the familiarization session if they are unable to perform the tasks or follow instructions, or if their TMS stimulation parameters cannot be reliably determined by the experimenter, or if TMS is not well tolerated.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Bloomington, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited with flyers posted in the community. They were asked to complete an electronic screening form to determine basic eligibility and, if they appeared eligible, the experimenter scheduled the familiarization session.
Pre-assignment Details: During the familiarization session, after giving informed consent, participants experienced the transcranial magnetic stimulation (TMS) used in the main experiment. This was to make sure they were not bothered by the sensations before random group assignment. Of the 118 who enrolled, 25 found the TMS uncomfortable and were excluded. A further 6 withdrew due to scheduling conflicts, leaving 87 who received a group assignment.
Period: Overall Study
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Supramarginal Gyrus (SMG) | Sham Control Group
Started | 29 | 28 | 30
Completed | 27 | 26 | 26
Not Completed | 2 | 2 | 4
Not completed — Withdrawal by Subject | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: These are the participants who did the main session, where baseline measurements were made.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Supramarginal Gyrus (SMG) | Sham Control Group | Total
Number analyzed (Participants) | 27 | 26 | 26 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (7.0) | 22.5 (3.6) | 23.1 (4.2) | 23.6 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 12 | 42
  Male | 13 | 10 | 14 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 4 | 14
  Not Hispanic or Latino | 24 | 19 | 22 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 12 | 11 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 14 | 11 | 12 | 37
  More than one race | 3 | 2 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 26 | 79
Edinburgh handedness inventory [Mean (Standard Deviation); unit: units on a scale] — Questionnaire to assess handedness. The scale ranges from -100 (fully left handed) to 100 (fully right handed).
  units on a scale | 89.2 (10.7) | 85.2 (16.5) | 78.4 (18.9) | 84.3 (16.1)
Resting Motor Threshold (RMT) [Mean (Standard Deviation); unit: Percent of max stimulator output (%MSO)] — TMS measure that reflects each person's motor cortex excitability. Used to determine the theta burst stimulation intensity for that individual.
  Percent of max stimulator output (%MSO) | 49.3 (9.7) | 50.7 (8.6) | 50.3 (8.0) | 50.1 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Motor Skill
Description: Assessed by measuring movement accuracy on a maze-tracing task. Accuracy is defined by percent of movement path that falls within the maze. Participants traced the maze 10 times at 3 different speed ranges. Overall performance accuracy was taken as the mean accuracy across the three speed ranges. A change in mean accuracy reflects learning.
Time Frame: Assessed 4 times during the 2-hour main session: Pre-cTBS ("Pre"), immediately post-cTBS ("Post1"), after 40 trials of maze-tracing practice ("Post2"), and after 80 trials of maze-tracing practice ("Post 3").
Measure: Mean (Standard Deviation); unit: Accuracy (%)
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Supramarginal Gyrus (SMG) | Sham Control Group
Number analyzed (Participants) | 27 | 26 | 26
Accuracy (%)
  Pre timepoint | 66.6 (9.3) | 59.4 (8.9) | 59.9 (10.6)
  Post 1 timepoint | 64.9 (10.5) | 58.5 (9.7) | 63.5 (9.1)
  Post 2 timepoint | 69.4 (8.6) | 61.8 (8.7) | 65.4 (10.9)
  Post 3 timepoint | 68.2 (11.6) | 62.1 (10) | 66.3 (11.3)
Statistical Analysis 1: Comparison: Dorsolateral Prefrontal Cortex (DLPFC) vs Sham Control Group; Test type: Superiority; p = 0.55, t-test, 2 sided — Pairwise p-values were calculated using independent-samples t-tests on final values because model-based pairwise contrasts were not available. These values do not reflect the full repeated-measures mixed-model structure; Mean Difference (Final Values) = 1.9
Statistical Analysis 2: Comparison: Supramarginal Gyrus (SMG) vs Sham Control Group; Test type: Superiority; p = 0.18, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.2

2. Primary Outcome: Proprioception
Description: Two-alternative forced choice task where the robot moves the participant's hand in two different positions, and the participant reports whether second position was closer or further than first position. This data is fitted with a logistic regression relating the distance between the two positions and the likelihood that participant reports "further". The outcome measure is the distance at which the participant is equally likely to say "closer" or "further"; this is defined as the point of subjective equality, which indexes proprioceptive accuracy. If the number is small (close to zero), it means the person has high proprioceptive accuracy. If the number is large, it means the person is less accurate.
Time Frame: Assessed at 2 timepoints during the 2-hour main session: pre-cTBS ("Pre") and post-cTBS ("Post").
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Supramarginal Gyrus (SMG) | Sham Control Group
Number analyzed (Participants) | 27 | 26 | 26
mm
  Pre timepoint | 0.9 (0.62) | 0.79 (0.72) | 0.73 (0.56)
  Post timepoint | 1.2 (1.14) | 0.8 (0.55) | 0.75 (0.79)
Statistical Analysis 1: Comparison: Dorsolateral Prefrontal Cortex (DLPFC) vs Sham Control Group; Test type: Superiority; p = 0.1, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.45
Statistical Analysis 2: Comparison: Supramarginal Gyrus (SMG) vs Sham Control Group; Test type: Superiority; p = 0.79, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.05

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during each study visit: the familiarization session (about 1 hour), the MRI (about 30 minutes), and the main session (about 2 hours).
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Supramarginal Gyrus (SMG) | Sham Control Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 5/28 | 7/28 | 6/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dorsolateral Prefrontal Cortex (DLPFC) (N=28) | Supramarginal Gyrus (SMG) (N=28) | Sham Control Group (N=30)
Discomfort from TMS (General disorders) | 4 (4) | 7 (7) | 5 (5)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Fatigue is known to impair task performance and motor skill learning. Each participant took approximately 2 hours to complete the main session, which could have resulted in fatigue and poor attention during or by the end of it, even with breaks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT05739994/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT05739994/ICF_001.pdf